CLINICAL TRIAL: NCT02173340
Title: Population Pharmacodynamic Modeling of the Sedative and Side Effects of Propofol in Patients Undergoing Spinal Anesthesia
Brief Title: Population Pharmacodynamic Modeling of the Sedative and Side Effects of Propofol
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 3-2011-0247
Record Dates: First submitted 2014-05-19; First posted 2014-06-24 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Surgery Related to Lower Extremity Under Spinal Anesthesia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Sedation during spinal anesthesia is very useful for patients' comfort. However, intermittent bolus of sedative frequently results in inappropriate sedation which comes with various side effects such as patients' discomfort and apnea. Therefore, it would be reasonable to use target-controlled infusion(TCI) to provide proper sedation without serious side effects.

In this study, the investigators try to find the appropriate propofol target concentration with TCI device and build a pharmacodynamic non-linear mixed effect model between propofol target concentration and side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients who have lower extremity surgery under spinal anesthesia and who want to be sedated

Exclusion Criteria:

* patients who have deafness, neurologic deficit, Glasgow coma scale less than 15, history of drug allergy and who are on central nervous system-related drugs,

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have lower extremity surgery under spinal anesthesia at Gangnam Severance Hospital
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
sedation score | every 5 minutes when the dose is adjusted up to 1 hour
  Sedation score will be assessed with 'Modified Observer's assessment of alertness/sedation (OAA/S) score'. It has 5 scales from 1 to 5 as followed.
  1. responds readily to name spoken in normal tone
  2. lethargic response to name spoken in normal tone
  3. responds only after name is spoken loudly and/or repeatedly
  4. responds only after mild prodding or shaking
  5. does not respond to mild prodding or shaking
  After induction of spinal anesthesia, patient will be sedated with propofol via TCI device. The infusion dose will be adjusted every 5 minutes until the OAA/S score reaches 4. The patient's OAA/S score will be assessed overtime the infusion dose is adjusted during sedation. At the same time, airway obstruction score will be assessed and if the score reaches 4, the dose will be reduced.

SECONDARY OUTCOMES:
airway obstruction score | every 5 minutes when the dose is adjusted up to 1 hour
  Airway obstruction score will be assessed as followed.
  1. normal breathing
  2. deep breathing
  3. snoring
  4. severe airway obstruction
  After induction of spinal anesthesia, patient will be sedated with propofol via TCI device. The infusion dose will be adjusted every 5 minutes until the OAA/S score reaches 4. The patient's OAA/S score will be assessed overtime the infusion dose is adjusted during sedation. At the same time, airway obstruction score will be assessed and if the score reaches 4, the dose will be reduced.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Woo Han, MD, PhD, Principal Investigator — Yonsei University Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea